CLINICAL TRIAL: NCT01256879
Title: Evaluation of Excipient Effects on Biopharmaceuticals Classification System (BCS) Class 3 Drug Cimetidine
Brief Title: Cimetidine Biowaivers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00046139; HHSF2232000910020C (Other Grant/Funding Number: HHSF2232000910020C)
Record Dates: First submitted 2010-11-15; First posted 2010-12-09 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: cimetidine; pharmacokinetics; formulation
MeSH Terms: interventions — Cimetidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CimTest-A (Experimental): 200mg cimetidine (as 2 capsules)
  Interventions: Drug: Drug: cimetidine
- CimTest-B (Experimental): 200mg cimetidine (as 2 capsules)
  Interventions: Drug: Drug: cimetidine
- Sorbitol-free cimetidine solution (Active Comparator): 200mg cimetidine (as oral liquid)
  Interventions: Drug: Drug: cimetidine
- Commercial cimetidine solution (Experimental): 200mg cimetidine (as oral liquid)
  Interventions: Drug: Drug: cimetidine

INTERVENTIONS:
Drug: Drug: cimetidine — cimetidine 200mg total dose (single dose) as either CimTest-A capsules, CimTest-B capsules, sorbitol-free solution, or commercial cimetidine solution
  Other Names: Tagamet

SUMMARY:
The purpose of this research is to see if non-drug ingredients in capsules and oral solutions affect how well drugs are absorbed. This is called "bioequivalence." Medications taken by mouth, such as capsules and solutions, need to be absorbed into the body in order to do any good. Capsules and solutions contain a drug, but also contain non-drug ingredients that are called excipients or fillers. Excipients in the capsules and solutions can impact how much drug is absorbed into the body. This is called "bioINequivalence." Capsules and solutions in this research contain the drug cimetidine. This drug is being used since it has high water solubility (can dissolve in water) and low ability to be absorbed.

DETAILED DESCRIPTION:
The investigators anticipate that common excipients do not cause bioINequivalence. 1) The hypothesize is that commonly used excipients in oral medications change the rate or extent of Class 3 drug absorption and result in bioINequivalence. 2) Alternative hypothesis is that commonly used excipients in oral medications do not change the rate or extent of Class 3 drug absorption and do not result in bioINequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 18-55
* Healthy volunteers: Subjects in good health, as determined by screening evaluation that is not greater than 30 days before the first drug study visit
* Willing to avoid caffeine containing products 24 hours prior to and day of study visits
* Willing to stop all over the counter medications for 24 hours prior to and during study visits
* Able to provide informed consent

Exclusion Criteria:

* Presence of significant medical disease (including cardiovascular, pulmonary, hematologic, endocrine, immunologic, neurologic, gastrointestinal or psychiatric)
* Presence of hepatic, renal disease
* Pregnant women, breast feeding or trying to become pregnant
* Excessive alcohol use (i.e. current physical, behavioral, or personal manifestations related to the abuse or dependency on alcohol)
* Routine use (i.e. daily or weekly) prescription medication except birth control pills
* Routine use (i.e. daily or weekly) use of acid blockers, antacids, anti-diarrhea, stimulants, appetite suppressants, or anti nausea medication or other drugs that modulate gastrointestinal function
* Currently taking cimetidine or medication known to interact with cimetidine
* Allergic to cimetidine
* Undergoing therapy for solid tumor or blood malignancy
* Any condition in which in the opinion of the PI or medical physician would increase risk to the subject or interfere with the integrity of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Polli, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Rege BD, Yu LX, Hussain AS, Polli JE. Effect of common excipients on Caco-2 transport of low-permeability drugs. J Pharm Sci. 2001 Nov;90(11):1776-86. doi: 10.1002/jps.1127. PMID 11745735

RESULTS

PARTICIPANT FLOW:
Groups:
- Cimetidine: cimetidine 200mg total dose (single dose)
Period: Overall Study
Arm/Group | Cimetidine
Started | 25 (25 started in this cross-over study but only 24 completed)
CimTest-A | 25 (25 started this intervention but only 24 completed)
CimTest-B | 24 (24 started this intervention and 24 completed)
Sorbitol-free Cimetidine Solution | 24 (24 started this intervention and 24 completed)
Commercial Cimetidine Solution | 24 (24 started this intervention and 24 completed)
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: healthy subjects
Arm/Group | Cimetidine
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: pharmacokinetic exposure (ng*hr/ml)
Time Frame: 0-10 hours
Measure: Mean (Standard Error); unit: ng*hr/ml
Groups:
- Experimental: CimTest-A: cimetidine capsule with hydroxypropyl methylcellulose (HPMC), a type of filler
  cimetidine: cimetidine 200mg total dose (single dose)
- Experimental: CimTest-B: cimetidine capsule with magnesium stearate, a type of filler
  cimetidine: cimetidine 200mg total dose (single dose)
- Active Comparator: Sorbitol-free Cimetidine Solution: non-commercial cimetidine solution
  cimetidine: cimetidine 200mg total dose (single dose)
- Experimental: Commercial Cimetidine Solution: commercial cimetidine solution
  cimetidine: cimetidine 200mg total dose (single dose)
Arm/Group | Experimental: CimTest-A | Experimental: CimTest-B | Active Comparator: Sorbitol-free Cimetidine Solution | Experimental: Commercial Cimetidine Solution
Number analyzed (Participants) | 24 | 24 | 24 | 24
ng*hr/ml | 3896 (181) | 3661 (186) | 3495 (183) | 3512 (193)
Statistical Analysis 1: Comparison: Experimental: CimTest-A vs Experimental: CimTest-B vs Experimental: Commercial Cimetidine Solution; Test type: Other — Each CimTest-A, CimTest-B, and Commercial Cimetidine Solution are compared to Active Comparator (i.e. Sorbitol-free Cimetidine Solution), as a percentage of Active Comparator, per routine FDA bioequivalence testing of AUC; Bioequivalence testing of AUC, per FDA guidance, is applied. Each CimTest-A, CimTest-B, and Commercial Cimetidine Solution are compared to Active Comparator (i.e. Sorbitol-free Cimetidine Solution), as a percentage of Active Comparator, per routine FDA bioequivalence testing of AUC. The upper and lower 90% Confidence Interval for CimTest-A is 104.4% to 120.6%. The upper and lower 90% Confidence Interval for CimTest-B is 97.9% to 113.0%. The upper and lower 90% Confidence Interval for Commercial Cimetidine Solution is 93.2% to 107.7%

ADVERSE EVENTS:
Time Frame: 10 hours
Arm/Group | Experimental: CimTest-A | Experimental: CimTest-B | Active Comparator: Sorbitol-free Cimetidine Solution | Experimental: Commercial Cimetidine Solution
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/25 | 0/24 | 0/24 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: CimTest-A (N=25) | Experimental: CimTest-B (N=24) | Active Comparator: Sorbitol-free Cimetidine Solution (N=24) | Experimental: Commercial Cimetidine Solution (N=24)
pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — pain at IV site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes